CLINICAL TRIAL: NCT00346463
Title: Does Antenatal Allopurinol Administration Improve Maternal and Neonatal Outcome in Intrauterine Growth Restriction?
Brief Title: Antenatal Allopurinol in Intrauterine Growth Restriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METC UMCU 05-207K
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2006-06

CONDITIONS: Fetal Growth Retardation
Keywords: Allopurinol; Fetal Growth Retardation; Oxidative Stress; Placental Insufficiency
MeSH Terms: conditions — Fetal Growth Retardation; Placental Insufficiency | interventions — Allopurinol

INTERVENTIONS:
Drug: Allopurinol

SUMMARY:
Growth retardation in utero may be caused by uteroplacental vascular insufficiency. When Doppler ultrasound studies of the umbilical artery are abnormal pathological intrauterine growth restriction (IUGR) can be diagnosed. IUGR fetuses have a higher mortality and morbidity, both perinatally and on the longer term. This is probably due to chronic malnourishment and hypoxia due to placental insufficiency. This placental dysfunction causes generation of harmful free oxygen radicals in the fetus. The IUGR fetus has a diminished antioxidative capacity which means these free radicals cannot be buffered sufficiently. This leads to fetal oxidative stress.

Previous studies have shown that allopurinol can inhibit the cascades that lead to generation of free radicals. High dosed allopurinol also scavenges radicals and binds free iron without adverse effects on the fetus or mother.

As IUGR is associated with placental insufficiency and excessive production of free radicals we hypothesize that antenatal allopurinol administration could lead to a decrease in oxidative stress in the mother and fetus and subsequent improvement of the maternal and/or neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

Mothers with a gestational age (GA) of 30 to 36 weeks with:

* Foetal growth retardation (growth <10th percentile) and
* Abnormal Doppler flow in the umbilical cord (umbilical artery pulsatility index (PI)>95th percentile)

Exclusion Criteria:

* Congenital, chromosomal or syndromal abnormalities
* Positive screening for intrauterine viral infections
* Mothers with gout and high uric acid
* creatinine > 100 umol/l
* ASAT > 80 U/l, ALAT > 80 U/l
* Uric acid > 0,50 mmol/l

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
free radical production / oxidative stress

SECONDARY OUTCOMES:
foetal parameters (Doppler, cardiotocography)
postponement of birth
morbidity (including long term neurodevelopmental outcome)
mortality
pharmacokinetices

CONTACTS AND LOCATIONS:
Overall Officials: Frank van Bel, Prof MD, PhD, Study Director — Wilhelmina Children's Hospital / UMC Utrecht; Manon Benders, MD, PhD, Principal Investigator — Wilhelmina Children's Hospital, UMC Utrecht; Helen Torrance, MD, Principal Investigator — Wilhelmina Children's Hospital / UMC Utrecht
Locations (1):
- Wilhelmina Children's Hospital / UMC Utrecht, Utrecht, Utrecht, Netherlands